CLINICAL TRIAL: NCT02423967
Title: A Comparison of Efficacy of Fresh Versus Frozen Donor Stool for Fecal Microbial Transplant in Children With Recurrent Clostridium Difficile Infections
Brief Title: Fresh Versus Frozen Stool for Fecal Transplant in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark G. Bartlett, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-004472
Record Dates: First submitted 2015-04-06; First posted 2015-04-22 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Clostridium Difficile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transplant uses fresh familial stool (Active Comparator): Undergoes Fecal Microbial Transplant using fresh stool from a screened family member Followed up and assessed for eradication of Clostridium difficile Quality of life assessed Stool assessed for inflammation and microbiome
  Interventions: Biological: Transplant uses fresh familial stool
- Transplant uses frozen anonymous stool (Experimental): Undergoes Fecal Microbial Transplant using stool collected from screened anonymous donor that has been frozen until time of Fecal Microbial Transplant Followed up and assessed for eradication of Clostridium difficile Quality of life assessed Stool assessed for inflammation and microbiome
  Interventions: Biological: Transplant uses frozen anonymous stool

INTERVENTIONS:
Biological: Transplant uses frozen anonymous stool — The intervention is using frozen anonymous donor stool instead of fresh stool from family members for the fecal microbial transplant to treat recurrent CDI.
  Other Names: fecal microbial transplant
  Arms: Transplant uses frozen anonymous stool
Biological: Transplant uses fresh familial stool — The intervention is using fresh familial donor stool for the fecal microbial transplant to treat recurrent CDI
  Other Names: fecal microbila transplant
  Arms: Transplant uses fresh familial stool

SUMMARY:
The primary goal of this study will be to assess whether stool collected and frozen from anonymous screened unrelated donors can be as effective as stool freshly collected from recipient's parents when used in Fecal Microbial Transplant for the eradication of recurrent Clostridium difficile infections in children. In the current protocols, which are more than 90% effective, each child who is receiving a fecal transplant has to provide their own donor stool, usually from a parent or close relative. This requires considerable screening costs for each case and is logistically complicated as the donor must be present and must stool just prior to the transplant. The investigators hope to show that a small number of healthy donors can provide stool samples which can be frozen and banked and then thawed for use in numerous patients. The primary goal is to show that Clostridium difficile will be eradicated as effectively (Greater than 90% success) when using the stool from the frozen donors.

The study will also evaluate the inflammatory response and intestinal microbiome in young children aged 1-3 years with Clostridium difficile infections to better predict which ones will respond to fecal transplantation and which ones have incidental infections. For this question the investigators will gather stool samples to check for lactoferrin, calprotectin, and alpha1antitrypsin, and 16s ribosomal RNA analysis in children before and after the fecal transplants. The goal is to see if there is an intestinal microbiome that predisposes some children to getting sick from Clostridium difficile versus just having it incidentally.

DETAILED DESCRIPTION:
The study is designed to enroll forty children aged 1-18 with recurrent Clostridium difficile Infection (CDI). Recurrent CDI is defined as an infection that persists after three rounds of appropriate antibiotics. Enrollees will be randomly assigned to receive Fecal Microbial Transplant using stool from either a screened relative as per current protocols versus using frozen stool that has been collected from healthy volunteers.

Primary outcome will be the eradication of the Clostridium difficile as defined by elimination of diarrhea with a negative Clostridium difficile toxin stool test.

Secondary outcomes will include a measure of quality of life pre and post Fecal Microbial Transplant using a validated quality of life survey instrument, the Health Act Child Health Questionnaire. The investigators will also assess for inflammation in the stool using lactoferrin and calprotectin and evaluate the stool microbiome in recipients pre and post transplant using sequencing to look for any pattern that predicts successful eradication.

ELIGIBILITY:
Eligible children between aged 1 and 18 years must have had Clostridium difficile infection that has not been eradicated despite at least two courses of antibiotics ( either metronidazole or vancomycin).

Inclusion criteria:

* Age 1-18 years
* Diarrhea
* Positive Clostridium difficile infection using stool toxin testing
* Diarrhea that has improved on antibiotics but recurs when antibiotics are stopped.
* Willingness to undergo Fecal Microbial Transplant using frozen stool from anonymous screened donors.

Exclusion Criteria:

* Age under 1 or over 18
* No diarrhea

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2015-04; Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Clostridium difficile (CD) Eradication; percentage of patients with negative CD toxin in stool following Fecal Microbiota Transplant | 4 weeks
  Will analyze stool sample collected 4 weeks after fecal microbiota transplant (FMT) for presence or absence of Clostridium difficile toxin. In addition, will note whether presenting symptoms improved or not after FMT.

SECONDARY OUTCOMES:
Changes in quality of life questionnaire scores after Fecal Microbiota Transplant | 12 weeks
  Will assess quality of life using standardized Child health Questionnaire which provides a raw score of 0-100. Investigators will compare scores of all patients before Fecal Transplant and 12 weeks after in order to mark the impact of procedure outcome on children's physical and psychological health
percentage of patients with stool Calprotectin levels exceeding 50 mcg/g after Fecal Microbiota Transplant | 4 weeks
  Will assess fecal Calprotectin levels in stools prior to fecal transplant and 4 weeks after
percentage of patients with positive Lactoferrin inflammatory marker in stools after Fecal Microbiota Transplant | 4 weeks
  Analyze stool samples for presence or absence Lactoferrin before Fecal transplant and 4 weeks after

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bartlett, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials